CLINICAL TRIAL: NCT06830707
Title: Effect of Lower Limb Constraint Induced Movement Therapy Using a Torque-Assisted Exoskeletal Wearable Device on Ambulatory Function in Late Subacute and Chronic Stroke Patients, Single-Center, Single-blinded Cross-over Prospective Pilot Study
Brief Title: Effect of Lower Limb Constraint Induced Movement Therapy Using a Torque-Assisted Exoskeletal Wearable Device
Acronym: CIMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Hyuk Chang, professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2022-07-088
Record Dates: First submitted 2025-01-13; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Chronic Stroke; Subacute Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Torque-Assisted Exoskeletal Wearable Device group (Experimental): The treatment comprised 5 robot-assisted gait training sessions over a 2-week period, followed by 10 lower limb Constraint Induced Movement Therapy(CIMT) sessions with a torque assisted exoskeleton.
  Interventions: Device: experimental group

INTERVENTIONS:
Device: experimental group — The treatment comprised 5 robot-assisted gait training sessions over a 2-week period, followed by 10 lower limb Constraint Induced Movement Therapy(CIMT) sessions with a torque assisted exoskeleton.

SUMMARY:
The aim of this study was to investigate the effects of lower limb constraint induced motor therapy using the robotic rehabilitation device on ambulatory function in chronic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older
* Patients with hemiparesis due to ischemic or hemorrhagic stroke
* Patients in the late subacute or chronic phase, at least 3 months after the onset of stroke
* Individuals who can independently walk with a Functional Ambulatory Category score of 3 or higher
* Patients who are able to use Torque-Assisted Exoskeletal Wearable Device Height: 140 cm to 190 cm Weight: 80 kg or less Shoe size: 230 mm to 290 mm
* Patients who were independent walkers and had no difficulties performing activities of daily living (mRS ≤ 1)

Exclusion Criteria:

* Patients with severe cognitive impairment (MMSE <10) or significant communication difficulties such as speech disorders
* Patients with spasticity in one-sided lower limbs, rated 2 or higher on the Modified Ashworth Scale (MAS)
* Patients with severe musculoskeletal disorders of the lower limbs
* Patients with contractures that limit the range of motion in the lower limbs
* Patients with an apparent leg length discrepancy of 2 cm or more
* Patients with fractures, open trauma, or non-healing ulcers in the lower limbs
* Patients with serious internal diseases such as cardiovascular disease or pulmonary disease that make it difficult to use Exoskeletal Wearable Device for walking therapy
* Patients with a history of osteoporotic fractures
* Patients with other neurological disorders affecting walking (e.g., Parkinson's disease, multiple sclerosis, etc.)
* Any other cases where the investigator determines that participation in this study is inappropriate

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Comparison of the change in walking speed | 3 weeks follow up
  Comparison of the change in walking speed before and after 5 sessions of walking training versus 10 sessions of CIMT exercise training

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea